CLINICAL TRIAL: NCT04567706
Title: Analysis of the Tumor Microenvironment and Immune Response in Malignant Melanoma
Brief Title: A Storage Facility for Tissues Obtained From Patients With Malignant Melanoma
Status: Recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, William Carson, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-13114; NCI-2020-06536 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-09-13; First posted 2020-09-28 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ancillary-correlative (biospecimen collection): Patients undergo collection of blood samples at the time of the initial diagnostic work-up, and possibly prior to the initiation of surgery, chemotherapy, immunotherapy, or radiation therapy, at tumor progression or recurrence, and annually during routine follow-up (no more than 4 blood draws per year). Patients may also undergo collection of tissue sample during standard of care surgical or radiologic procedures. Healthy individuals undergo collection of blood samples up to 4 times over 1 year.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and tissue samples

SUMMARY:
This study collects and stores blood and tumor samples from patients with malignant melanoma and healthy individuals. The purpose of this study is to gain a better understanding of the causes of melanoma and how melanoma tumors behave. Storing blood and tumor samples for future research may lead to new discoveries that may ultimately help with diagnosing or treating this disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Facilitate studies aimed at investigating new prognostic markers and potentially therapeutic therapies in malignant melanoma.

OUTLINE:

Patients undergo collection of blood samples at the time of the initial diagnostic work-up, and possibly prior to the initiation of surgery, chemotherapy, immunotherapy, or radiation therapy, at tumor progression or recurrence, and annually during routine follow-up (no more than 4 blood draws per year). Patients may also undergo collection of tissue sample during standard of care surgical or radiologic procedures. Healthy individuals undergo collection of blood samples up to 4 times over 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patient with malignant melanoma or personal history of melanoma
* Normal donors
* Informed consent can be obtained
* Patients with any stage of malignant melanoma

Exclusion Criteria:

* Incarcerated individuals will be excluded from this protocol

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are being evaluated or treated for malignant melanoma by members of the departments of Surgical Oncology, Medical Oncology, and Radiation Oncology and normal controls
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-05-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
New prognostic markers in malignant melanoma | Up to 3 months
  Facilitate studies aimed at investigating new prognostic markers and potentially therapeutic therapies in malignant melanoma. . Draws conducted at baseline prior to immune therapy, four weeks after draw 1 and prior to the third cycle.

CONTACTS AND LOCATIONS:
Overall Officials: William E Carson, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu